CLINICAL TRIAL: NCT05767242
Title: Early Neurophysiological Markers of Language Impairments: a Longitudinal Study on Infants At Familial Risk
Brief Title: Early Neurophysiological Markers of Language Impairments
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 918
Record Dates: First submitted 2023-01-26; First posted 2023-03-14 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Development, Infant; Development, Language; Developmental Language Disorder; Learning Disabilities
MeSH Terms: conditions — Language; Language Development Disorders; Learning Disabilities | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MEDEA BabyLab Cohort
  Interventions: Other: Electrophysiological recording; Behavioral: Behavioral assessment

INTERVENTIONS:
Other: Electrophysiological recording — Investigation of early neural markers using electrophysiology at 6-12-24 months
Behavioral: Behavioral assessment — Individual behavioral assessment at later ages (3, 4.5, 6, and 8 years)

SUMMARY:
The present project aims at identifying very early electrophysiological risk markers for language impairments. The long-term goals of the study include the characterization of learning developmental trajectories in children at high risk for language impairments. In this project, all the infants of the Medea BabyLab cohort are followed-up until school age. Since these infants have complete information on early electrophysiological markers, the final goal of the project is the characterization of their learning developmental trajectories and the construction of a multi-factor prognostic model that includes the neurophysiological processes underlying basic-level skills as potential biomarkers for predicting later reading and spelling skills.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged <24 months
* Infants with and without familial risk for language impairments (infants are assigned to the group with familial risk if at least one first-degree relative had a certified (clinical) diagnosis of language impairment or learning disability
* Both parents are native-Italian speakers

Exclusion Criteria:

* Gestational age < 37 weeks and/or birth weight < 2500 grams
* APGAR scores at birth at 1' and 5' < 7
* Bayley Cognitive Score < 7
* Presence of certified diagnosis of intellectual deficiency, attention-deficit disorder, sensorial and neurological disorders, or autism within first-degree relative

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants with and without familial risk for language impairments
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Expressive vocabulary at age 3 years | Age 3 years
  Standardized score in the Language Development Survey (Rescorla, 1989; Rescorla et al., 2014). Minimum=5; Maximum=95 (higher scores mean a better outcome).
Phonological awareness at age 3 years | Age 3 years
  Raw score in a syllabic blending task (created ad hoc). Scores are percentages of accuracy (higher scores mean a better outcome).
Syntactic comprehension at age 3 years | Age 3 years
  Standardized scores in the syntactic comprehension subtests, taken from 'Test for language evaluation', Cianchetti e Fancello, 1997. Z-scores are calculated (higher scores mean a better outcome).
Lexical comprehension at age 3 years | Age 3 years
  Raw score in the lexical comprehension subtest, taken from 'Battery for language evaluation in children 4-12 years', Marini et al., 2015. Scores are percentages of accuracy (higher scores mean a better outcome).
Short-term verbal memory at age 4.5 years | Age 4.5 years
  Standardized scores in the pseudo-word repetition subtest, taken from 'Battery for language evaluation in children 4-12 years', Marini et al., 2015. Z-scores are calculated (higher scores mean a better outcome).
Phonological awareness at age 4.5 years | Age 4.5 years
  Standardized scores in the phonological awareness subtests taken from 'Evaluation of phonological awareness skills', Marotta et al., 2008. Mean=10, Standard Deviation=3 (higher scores mean a better outcome).
Phonological awareness at age 6 years | Age 6 years
  Composite score of the standardized scores in the phonological awareness subtests (phoneme identification, phonemic segmentation), Cornoldi et al., 2009. Z-scores are calculated (higher scores mean a better outcome).
Letter identification, knowledge, and writing at age 6 years | Age 6 years
  Raw scores in the letter identification, knowledge, and writing subtests, taken from "Preschool Screening", Savelli et al., 2013. Minimum=0, Maximum=20 (higher scores mean a better outcome).
Reading (accuracy, speed and comprehension) at age 8 years | Age 8 years
  Standardized scores in the reading subtest, taken from 'Reading and comprehension assessment', Bonifacci et al., 2014. Z-scores are calculated (higher scores mean a better outcome).
Spelling at age 8 years | Age 8 years
  Standardized scores in the spelling task (Marinelli et al., 2016). Z-scores are calculated (higher scores mean a better outcome).
Phonemic awareness at age 8 years | Age 8 years
  Raw scores in the spoonerisms subtest taken from 'Evaluation of phonological awareness skills', Marotta et al., 2008. Minimum=0, Maximum=30 (higher scores mean a better outcome).

SECONDARY OUTCOMES:
Lexical access at age 4.5 years | Age 4.5 years
  Standardized score in Rapid Automatic Naming. Mean=10, Standard Deviation=3 (higher scores mean a better outcome).
Naming and articulatory accuracy at age 3 years | Age 3 years
  Raw scores in the test of naming and articulatory accuracy (created ad hoc). Scores are percentages of accuracy (higher scores mean a better outcome).
Nonverbal cognitive score at age 4.5 years | Age 4.5 years
  Standardized score in the block design subtest, taken from 'Wechsler Preschool and Primary Scale of Intelligence, 3rd edition'. Mean=10, Standard Deviation=3 (higher scores mean a better outcome).
Lexical access at age 6 years | Age 6 years
  Standardized score in Rapid Automatic Naming, taken from Urgesi et al., 2011. Z-scores are calculated (higher scores mean a better outcome).
Visual-motor integration at age 6 years | Age 6 years
  Standardized score in the 'Developmental Test of Visual-Motor Integration', Preda, 2000. Minimum=5; Maximum=95 (higher scores mean a better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Associazione La Nostra Famiglia - IRCCS Eugenio Medea, Bosisio Parini, LC, Italy

IPD SHARING:
Plan to Share IPD: No